CLINICAL TRIAL: NCT05030844
Title: The Effect of IMB Model-Based Diabetes Education and Motivational Interviewing on Care Outcomes in Adults With Type 2 Diabetes-A Randomized Controlled Study: Randomized Controlled Trial
Brief Title: The Effect of IMB Model-Based Diabetes Education and Motivational Interviewing on Care Outcomes in Adults With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, EDA KILINÇ, Research Assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EKILINC
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Type2 Diabetes; Self Efficacy; Self Management; HbA1c; BMI
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled study
Who Masked: Participant
Masking Description: Single blinding was provided that included inclusion criteria and agreement to participate in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): IMB model-based interventions were applied to the intervention group for 3 month. For the information component of the IMB model, diabetes education consisting of four sessions was given in groups of five in the first two weeks. Each patient was given a "Diabetes Management Education Booklet" prepared by the researchers. For the motivation component of the IMB model, total 5 sessions 30-minute motivational interview was made with individual Whatsapp calls once every two weeks starting from the third week.
  Interventions: Behavioral: IMB model based Diabetes Education and Motivational Interviewing
- Control Group (No Intervention): The control group received routine nursing care in the endocrine policlinic.

INTERVENTIONS:
Behavioral: IMB model based Diabetes Education and Motivational Interviewing — IMB model-based interventions were applied to the intervention group for 3 month. For the information component of the IMB model, diabetes education consisting of four sessions was given in groups of five in the first two weeks. Each patient was given a "Diabetes Management Education Booklet" prepared by the researchers. For the motivation component of the IMB model, total 5 sessions 30-minute motivational interview was made with individual Whatsapp calls once every two weeks starting from the third week.
  Arms: Intervention Group

SUMMARY:
This study was conducted to examine the effects of IMB model-based diabetes education and Motivational Interviewing for adults with Type 2 diabetes on care outcomes This study was conducted to examine the effects of IMB model-based diabetes education and Motivational Interviewing interventions on care outcomes for adults with Type 2 diabetes (diabetes knowledge, health belief, self-efficacy, self-management, HbA1c and BKİ).

DETAILED DESCRIPTION:
This study was conducted to examine the effects of Information, Motivation and Behavioral Skills (IMB) model-based diabetes education and motivational interviewing on care outcomes in adults with Type 2 diabetes. The study is a single-blind, randomized controlled trial with pre-test, post-test and follow-up test measurements from experimental research designs. The study was carried out in the Endocrinology and Metabolic Diseases Polyclinic, and the data were collected between June 2021 and February 2022. The sample of the study (intervention group=30, control group=30) consisted of 60 individuals with type 2 diabetes. Study data were collected with Adult Diabetes Information Scale, Health Belief Model Scale, Diabetes Self-Efficacy Scale, Diabetes Self-Management Scale and metabolic control parameters follow-up form. IMB model-based diabetes education and motivational interview program were applied to the individuals in the experimental group for three months. Initially, diabetes education was given in small groups in four sessions, then Motivational Interviews were held individually every two weeks for a total of five sessions via WhatsApp.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 30-64
* Receiving insulin therapy
* BMI value of 25 and above
* HbA1c of 7 and above
* At least primary school graduate and can speak Turkish
* No communication barrier (speech, vision or hearing problem)
* Having a smart phone and internet access
* Individuals who agree to participate in the research.

Exclusion Criteria:

* Those who have retinopathy at a level that may hinder the sense of sight.
* Those with neuropathy at a level that prevents them from doing their daily physical activities
* Diagnosed with kidney failure
* Using an insulin pump
* Pregnant
* Those with a diagnosis of cancer

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
The change in diabetes knowledge level of individuals with Type 2 diabetes at 3rd month and 6 rd month with the Diabetes Knowledge Scale. | baseline, 3rd month and 6 rd month
  This scale was used to measure the knowledge component in the IMB model of individuals. The scale was developed by Erener Yavuz and Erol (2019) to measure the knowledge level of adults with diabetes. The scale consists of 5 sub-dimensions, including General Information on Diabetes (6 items), Blood Glucose Measurements and Values (5 items), Diabetes Risk Factors (4 items), Diabetes Symptoms (8 items), Diabetes Complications (5 items), and 28 consists of matter. Scale answers consist of two sets of items, true and false. Among the yes/no/don't know answer type questions, 1 point is given to those who give correct answers, 0 points are given to those who do not know and give wrong answers. The maximum score that can be obtained from the scale is 28, and the minimum score is 0.
The change in diabetes health belief of individuals with Type 2 diabetes at 3rd month and 6 rd month with the Health Belief Model Scale in Diabetes Patients. | baseline, 3rd month and 6 rd month
  This scale was used to measure the individual motivation component in the IMB model of individuals. The scale consists of 5 sub-dimensions and 33 items: perceived sensitivity (4 items), perceived seriousness (3 items), perceived benefits (7 items), perceived barriers (9 items), recommended health-related activities (10 items). The mean score of each sub-dimension is determined by dividing the total scores of all items in the sub-dimension by the total number of items. The total scale mean score is calculated by dividing the total scores of all scale items by the total number of items. The minimum score for each item is 1 and the maximum score is 5. Rating was made as strongly disagree (1), strongly agree (5). Low scores indicate negative and high scores indicate positive health beliefs. If the mean score for each item is 4 and above, it indicates high or positive health belief, and if the mean score is less than 4, it indicates low health belief.
The change in diabetes self efficacy of individuals with Type 2 diabetes at 3rd month and 6 rd month with the Diabetes Self-Efficacy Scale. | baseline, 3rd month and 6 rd month
  The "Self-Efficacy Scale" for diabetes management in type 2 diabetes patients was developed to determine the perception of diabetes patients' own power to carry out their own care activities. The items that make up the scale are based on the following activities. Activities to be done for diabetes treatment (drug use, diet, physical exercise), self-monitoring, self-control (knowing the value of blood sugar, body weight, foot control, general health), regulating their own activities (hypoglycemia, hyperglycemia correction, preparing for vacation) change in diet, overweight, self-control in case of illness and stress). The scale consists of 20 items. The lowest score to be taken from the scale is 20, and the highest score is 100.
The change in diabetes self managament of individuals with Type 2 diabetes at 3rd month and 6 rd month with the Diabetes Self-Management Scale | baseline, 3rd month and 6 rd month
  This scale was used to measure the behavioral component of individuals in the IMB model. The validity and reliability study of the Turkish Diabetes Self-Management Perception Scale was conducted by Eroğlu and Sabuncu (2018). The scale consists of 16 items and 4 sub-dimensions and is a 4-point Likert type. Glucose Management sub-dimension: Items 4, 6, 10, 12 (items 4 and 12 are about drug use, items 1, 6 and 10 are about blood glucose monitoring). Diet Control sub-dimension: Items 2, 5, 9, 13. Physical Activity sub-dimension: Items 8, 11, 15. Use of Health Services sub-dimension: It consists of 3, 7, 14, and 16 items. The DMS scale consists of 16 items, 7 of which are straight and 9 of which are reversed. The scores of the items numbered "5, 7, 10, 11, 12, 13, 14, 15 and 16" in the scale are calculated by reversing them. Diabetes self-management increases as the score gets closer to 10.

SECONDARY OUTCOMES:
Metabolic control variables | baseline, 3rd month and 6 rd month
  Measurement of changes in HbA1c and Body Mass Index levels of individuals with Type 2 diabetes at 3rd month and 6 rd month

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilinc Isleyen E, Kartal A. The effect of information, motivation and behavioural skills model-based Diabetes Education and Motivational Interview Program on health outcomes in middle-aged adults with type 2 diabetes: a randomised controlled study. Psychogeriatrics. 2025 Jan;25(1):e13219. doi: 10.1111/psyg.13219. Epub 2024 Nov 19. PMID 39562051